CLINICAL TRIAL: NCT01496222
Title: The Montreal Cognitive Assessment as a Screening Tool for Preoperative Mild Cognitive
Brief Title: The Montreal Cognitive Assessment as a Screening Tool for Preoperative Mild Cognitive Impairment in Geriatric Patients
Acronym: MoCA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phongthara Vichitvejpaisal", Professor Dr., Mahidol University
Other Study IDs: 460/2554(EC2)
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; Montreal Cognitive Assessment test
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, double-blinded, control trial. The Montreal Cognitive Assessment is used to screen preoperative mild cognitive impairment in 582 consecutive geriatric patients, scheduled for general, vascular or urological surgery under general and/or regional anesthesia.

DETAILED DESCRIPTION:
At the preoperative visit, the co-researcher invites 322 general and vascular patients (male 190, female 132) and 260 urological patients (male 220, female 40) who meet the inclusion criteria to join the study. The process of the project is explained to the interested patients in details before an informed consent is obtained.

All participants are interviewed by using the Montreal Cognitive Assessment test. The history of drug used preoperatively (medication reconciliation) has also been recorded.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 65 yr, ASA I-III scheduled for elective general, vascular or urological surgery under general and/or regional anesthesia.

Exclusion Criteria:

* unable to communicate in reading and writing
* psychosomatic patients
* insulin-dependant diabetes
* renal insufficiency (creatinine >1.5 mg/dL), renal dialysis
* uncontrolled congestive heart failure (American Heart Association Classification III or IV congestive heart failure), unstable angina, untreated cardiac arrhythmia
* active gastrointestinal bleeding.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study enrolls 582 consecutive geriatric patients,322 general and vascular patients (male 190, female 132) and 260 urological patients (male 220, female 40) who undergoing general and/or regional anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of mild cognitive impairment in preoperative geriatric patients | 1 Year

SECONDARY OUTCOMES:
Relationship between mild cognitive impairment and drug used preoperatively in geriatric patients | 1 year
  Pearson correlation coefficient will be used to evaluate the relationship between mild cognitive impairment and drug used preoperatively in geriatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Phongthara Vichitvejpaisal, M.D., Ph.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand